CLINICAL TRIAL: NCT01957449
Title: Safety and Efficacy of Propranolol in Severely Burned Children
Brief Title: Propranolol in Severely Burned Children
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: At the request of the study site, this study has been closed and access to study-related data is unavailable. We are unable to submit the results-data.
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Shriners Hospitals for Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-103
Record Dates: First submitted 2013-09-04; First posted 2013-10-08 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2018-08

CONDITIONS: Burn
MeSH Terms: conditions — Burns | interventions — Propranolol; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propranolol (Active Comparator): Propranolol by mouth given daily throughout hospitalization for up to 12 months
  Interventions: Drug: Propranolol
- Sugar Pill (Placebo Comparator): Placebo by mouth given daily throughout hospitalization for up to 12 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — Propranolol by mouth given daily throughout hospitalization for up to 12 months
  Other Names: Metoprolol; inderal
  Arms: Propranolol
Drug: Placebo — Placebo by mouth given daily throughout hospitalization for up to 12 months.
  Other Names: Control
  Arms: Sugar Pill

SUMMARY:
To determine the safety and efficacy of administration of propranolol for reducing heart rate and blood pressure in burn injury.

DETAILED DESCRIPTION:
Other purposes of this study are to study the effect on muscle function, the infectious process, sepsis, systemic inflammation and long-term scarring. Quality of life will also be looked at over time.

ELIGIBILITY:
Inclusion Criteria:

* Burns covering >20% of the total body surface are
* Age of 0 to 18 years
* Patient arrival to the burn center within 96 hours (4 days) of burn injury
* Require > 1 surgical procedure

Exclusion Criteria:

* Pregnancy
* Known history of AIDS, Aids Related Complex, or HIV
* History of cancer within 5 years
* Existence of pre-morbid conditions
* Asthma
* Congestive heart failure (measured ejection fraction < 20%)
* Medical condition requiring glucocorticoid treatment
* Burn injury due to chemical burns
* Burn injury due to deep electrical injury (decision of hospital PI)
* Presence of anoxic brain injury that is not expected to result in complete recovery
* Decision not to treat due to burn injury severity

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-04-23 (Actual)

PRIMARY OUTCOMES:
Resting heart rate multiplied by the systolic blood pressure measurement= rate pressure product | Measured during acute hospital stay, an average of 4 weeks.
  Multiply the subjects resting heart rate and systolic blood pressure measurements and average every 24 hours while hospitalized (an average of 4 weeks)

SECONDARY OUTCOMES:
Number of deaths | time of randomization up to one year
  Number of deaths will be compared between placebo group and propranolol treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: David N Herndon, MD, Principal Investigator — University of Texas
Locations (4):
- United States (4):
  - Shriners Hospitals for Children, Sacramento, California
  - Shriners Hospitals for Children, Boston, Massachusetts
  - Shriners Hospitals for Children, Cincinnati, Ohio
  - Shriners Hospitals for Children, Galveston, Texas

IPD SHARING:
Plan to Share IPD: No